CLINICAL TRIAL: NCT03208543
Title: Effectiveness, Safety and Feasibility of Thermotherapy With the Hand-held Exothermic Crystallization Thermotherapy for Cutaneous Leishmaniasis (HECT-CL), Device for Cutaneous Leishmaniasis in Quetta, Pakistan
Brief Title: Effectiveness, Safety and Feasibility of HECT-CL, in Quetta, Pakistan
Acronym: HECT-CL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: failure rate 91.1%
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HECT-CLQTA
Record Dates: First submitted 2017-05-26; First posted 2017-07-05 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Cutaneous Leishmaniases
Keywords: thermotherapy; Pakistan
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Hyperthermia

STUDY DESIGN:
Intervention Model Description: Patients meeting inclusion criteria will be enrolled to receive seven treatment sessions with thermotherapy (HECT-CL device) and will be reassessed during follow up visits at day 15, 30, 60, 90 and 180
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HECT-CL (Experimental): HECT-CL heat pack will be applied on CL lesions (50-52 degrees Celsius for 3 minutes on 7 consecutive days)
  Interventions: Device: HECT-CL

INTERVENTIONS:
Device: HECT-CL — To evaluate the effectiveness, safety and feasibility of thermotherapy with the low cost Hand-held Exothermic Crystallization Thermotherapy pad in the treatment of cutaneous leishmaniasis in Quetta, Balochistan, Pakistan.

SUMMARY:
This research studies the effect thermotherapy as treatment of Old World CL which is not invasive, non-toxic, and the short treatment. While the current standard treatment comprise daily painful injections with antimonials,

DETAILED DESCRIPTION:
The current standard treatment for Old World CL is based on daily painful injections with antimonials, which in Pakistan requires specialised care provided in secondary level care facilities.

Apart from potential toxic side effects of these antimonials, the long treatment course, high cost and inconvenience, it may prevent patients from seeking care or completing treatment, especially women and children in the Pakistan context. Untreated cutaneous leishmaniasis may leave disfiguring scars leading to stigmatisation and (psycho) social problems. If the CL lesions/scars are located on joints they can cause problems in motion and lead to disability. At a public health level, patients with untreated CL lesions are a reservoir for further transmission of CL in the family and community.

Thermotherapy is topical, not invasive, non-toxic, and the treatment duration is only 7 days, and therefore is expected to have major benefits for patients.

Additional advantages are that the HECT-CL can be applied by lower level qualified health workers, and the costs are low (less than 3 USD) per re-usable heat pad), and therefore can be rolled out to peripheral health facilities, potentially having a major impact on access to treatment.

ELIGIBILITY:
Inclusion criteria

* Patients with clinical CL symptoms for less than 6 months with the diagnosis confirmed by microscopic visualisation of Leishmania parasites in skin scrape smear.
* Patients who have given written informed consent.

Exclusion criteria

* Patients presenting with CL lesions located on or within two centimetres of eyes and lips.
* Patients with more than four lesions.
* Lesions, nodules and/or ulcerations with a diameter (ø) of more than 6 cm.
* Patients with persistent lesions for more than 6 months.
* Patients younger than 10 years.
* Patients who are unlikely, unable or unwilling to be available for and comply to regular follow up visits for 6 months.
* Pregnant, and lactating women <6 months after delivery.
* Patients with uncontrolled medical illnesses.
* Patients with immune disorders, such as HIV/AIDS, or those who are on steroid medication

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the HECT-CL treatment as assessed by | 180 days
  The proportion of patients with complete re-epithelisation at each follow up visit associated with the HECT-CL treatment
Possible adverse effect of the HECT-CL treatment will studied by | 180 days
  The proportion of patients experiencing adverse effects (AEs) and serious adverse effects (SAEs) (Safety)
Ease of use of the HECT-CL treatment as assessed by | 180 days
  the observation of, and feedback from health providers on the ease of (re-)use of the HECT-CL (feasibility).
Acceptability of the HECT-CL treatment as assessed by | 180 days
  proportion of patients completing the treatment schedule in time (feasibility)
Inappropriateness of the HECT-CL treatment as assessed by | 180 days
  the percentage of patients (%) with lesions where HECT-CL cannot be used, (e.g. near eyes and lips, larger than 6 cm, or more than four lesions) (feasibility)

SECONDARY OUTCOMES:
The scars remaining after the HECT-CL treatment as assessed by | 180 days
  the proportion of patients with remaining scars
The duration of the healing process as assessed by | 180 days
  The mean time (days) between time of start of treatment and complete re-epithelisation of the treated lesion the healing of the lesion (time-to-heal).

CONTACTS AND LOCATIONS:
Overall Officials: Koert Ritmeijer, PhD, Study Director — Medecins Sans Frontieres, Netherlands
Locations (1):
- Mohtarma Shaheed Benazir Bhutto Hospital Quetta., Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shah SA, Memon AA, Auwj-e-Shamim, Baqi S, Witzig R. Low-cost thermotherapy for cutaneous leishmaniasis in Sindh, Pakistan. J Pak Med Assoc. 2014 Dec;64(12):1398-404. PMID 25842586
- [Background] Olliaro P, Vaillant M, Arana B, Grogl M, Modabber F, Magill A, Lapujade O, Buffet P, Alvar J. Methodology of clinical trials aimed at assessing interventions for cutaneous leishmaniasis. PLoS Negl Trop Dis. 2013;7(3):e2130. doi: 10.1371/journal.pntd.0002130. Epub 2013 Mar 21. PMID 23556016
- [Background] Reithinger R, Mohsen M, Wahid M, Bismullah M, Quinnell RJ, Davies CR, Kolaczinski J, David JR. Efficacy of thermotherapy to treat cutaneous leishmaniasis caused by Leishmania tropica in Kabul, Afghanistan: a randomized, controlled trial. Clin Infect Dis. 2005 Apr 15;40(8):1148-55. doi: 10.1086/428736. Epub 2005 Mar 16. PMID 15791515
- [Background] Valencia BM, Miller D, Witzig RS, Boggild AK, Llanos-Cuentas A. Novel low-cost thermotherapy for cutaneous leishmaniasis in Peru. PLoS Negl Trop Dis. 2013 May 2;7(5):e2196. doi: 10.1371/journal.pntd.0002196. Print 2013. PMID 23658851